CLINICAL TRIAL: NCT04156412
Title: AXONE-Acute II: Acute Assessment of a Micro Multipolar Lead for Enhanced Cardiac Resynchronisation Therapy
Acronym: AXONE-Acute-2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Rouen (Other)
Collaborators: MicroPort CRM (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2019/127/HP
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Cardiac Resynchronisation Therapy
Keywords: quadripolar LV leads

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Implant test procedure (Experimental): Implant test procedure with new LV quadripolar lead before a standard implantation for Cardiac resynchronisation therapy
  Interventions: Device: Implant test procedure

INTERVENTIONS:
Device: Implant test procedure — Implant test procedure with new LV quadripolar lead before a standard implantation for Cardiac resynchronisation therapy

SUMMARY:
Pilot study to evaluate the performance of a lead below 2 French with specific distal shape to deliver efficient LV pacing

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient aged ≥18 years old.
* Patient presenting a CRT-P or CRT-D indication according to the latest ESC guidelines1.
* Primary implant of a CRT device (including upgrade from a single or dual-chamber pacemaker or ICD).
* Signed and dated informed consent.

Exclusion Criteria:

* Class IV of NYHA (ambulatory or not).
* Allergy to contrast media used for imaging during cardiac catheterization.
* Severe Renal Failure (clearance of creatinine according to Modification of diet in renal disease formula (MDRD) < 30ml/mn/m²).
* Previous failure of catheterization of the coronary sinus, or previous failure of left ventricular lead implantation.
* Already included in another clinical study involving intra-cardiac active implantable device, or participation to any other clinical trial in the last 2 weeks.
* Vulnerable patient such as person deprived of liberty by administrative or judicial decision or placed under judicial protection (guardianship or supervision).
* Known pregnancy, breastfeeding or women in childbearing age without an adequate contraceptive method with a known failure rate < 1%.-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-01-02 (Actual); Primary Completion 2020-09-29 (Actual); Study Completion 2020-09-29 (Actual)

PRIMARY OUTCOMES:
LV Bi-zone pacing success rate | 30 min
  Percent of patients where the placement of the AXONE lead provides two distant LV pacing vectors matching: Pacing Threshold ≤ 3.5V/0.5ms.
LV pacing success rate | 30 min
  Percent of patients where the placement of the AXONE lead allows at least one LV pacing vectors matching: Pacing Threshold ≤ 3.5V/0.5ms.

SECONDARY OUTCOMES:
Device or Implant testing procedure-related Adverse Events | 1 month post intervention
Electrical performance (1) | 30 min
  LV pacing threshold (Volt)
Electrical performance (2) | 30 min
  LV pacing impedance (Ohm)
AXONE Implant Efficiency (1) | 30 min
  procedure time for successful placement
AXONE Implant Efficiency (2) | 30 min
  fluoroscopic time
AXONE Implant Efficiency (3) | 30 min
  radiation dose
AXONE Implant Efficiency (4) | 30 min
  handling assessment.
LV multipoint pacing success | 30 min
  the placement of the AXONE provides two pacing vectors matching

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric ANSELME, Pr, Principal Investigator — University Hospital, Rouen
Locations (7):
- France (5):
  - Bordeaux University Hospital, Bordeaux
  - Clermont-Ferrand University Hospital, Clermont-Ferrand
  - Lille University Hospital, Lille
  - Rennes University Hospital, Rennes
  - Rouen University Hospital, Rouen
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Universitario y Politécnico La Fe, Valencia

IPD SHARING:
Plan to Share IPD: No